CLINICAL TRIAL: NCT03478540
Title: Impact of Gut Microbiota on the Immune Recovery in HIV-infection
Brief Title: Gut Microbiota and Immune Recovery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, Vice Director, Shanghai Public Health Clinical Center
Other Study IDs: Mic-1
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Anti-Retroviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-Retroviral Agents — First line antiretroviral therapy as recommended in China, e.g. tenofovir lamivudine and efavirenz

SUMMARY:
To explore whether gut microbiota would impact CD4 T cells recovery in HIV-infected patients on antiretroviral therapy (ART). We prospectively enroll patients initiate ART and collect their fecal at followup for one year.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Antiretroviral therapy naive
* CD4 T cell counts<350cells/mm3
* Agree to participate

Exclusion Criteria:

* Don't want to start antiretroviral therapy
* Cocurrent cancer or opportunistic infection
* Liver diseases
* received antibiotics within four weeks of enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected patients initiating antiretroviral therapy with CD4 T cell counts< 350cells/mm3
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Immune recovery | 48 weeks
  Cluster of differentiation 4 (CD4) T cells increased >25% or to higher than 350 cells/mm3

SECONDARY OUTCOMES:
HIV viral load | 48 weeks
  Viral load below limitation of detection
Microbiota composition | week 0 and 48
  Gut microbiota composition

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No